CLINICAL TRIAL: NCT04006392
Title: A Double-blind, Placebo-controlled Randomized Evaluation of the Effect of the Erchonia® FX-635™ on Diabetic Peripheral Neuropathy Pain
Brief Title: An Evaluation of the Effect of Low Level Laser Therapy on Diabetic Peripheral Neuropathy Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC_DPN2
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Erchonia FX-635 (Experimental): The Erchonia FX-635 is administered to the foot 12 times over 6 weeks (2 times each week) for 15 minutes per foot.
  Interventions: Device: Erchonia FX-635
- Placebo Laser (Sham Comparator): Noise and appearance of output is the same but no active therapy applied. Treatment administration procedure is the same as with the experimental arm.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia FX-635 — The Erchonia FX-635 has three independent 17 milliWatts (mW) 635 nanometer (nm) red laser diodes mounted in scanner devices.
  Arms: Erchonia FX-635
Device: Placebo Laser — Non-therapeutic output.
  Arms: Placebo Laser

SUMMARY:
The purpose of this study is to determine whether low level laser therapy is effective in the reduction of foot pain associated with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Peripheral neuropathy is one of the most common chronic diseases and a leading cause of adult disability in the U.S. Diabetic neuropathy represents over a third of all neuropathies, making diabetes the leading cause of peripheral neuropathy, affecting about 15-18 million Americans.

Living with neuropathy can cause tremendous frustration and social isolation. The daily chronic pain impacts day-to-day functionality resulting in physical and psychological problems including impaired concentration, anxiety, depression, a decline in cognitive abilities, and sleep difficulties which in turn can lead to irritability and increased pain sensitivity. Additionally, the economic burden from medical costs and workplace productivity losses are high and on the rise as the incidence of peripheral neuropathy increases.

Peripheral neuropathy describes damage to the peripheral nervous system that interferes with vital nerve connections, distorting and sometimes interrupting messages between the brain and the rest of the body. Diabetic peripheral neuropathy is a chronic acquired form of nerve damage that can occur in individuals with diabetes wherein the primary cause is damage to nerve fibers and blood vessels from prolonged exposure to high blood sugar (glucose). While the precise mechanism for this damage remains unclear, a combination of factors likely plays a role, including the complex interaction between nerves and blood vessels. High blood glucose interferes with the ability of the nerves to transmit signals and weakens the walls of the small blood vessels (capillaries) that supply the nerves with oxygen and nutrients.

The primary and most debilitating symptom of diabetic peripheral neuropathy is a sensation of tingling, prickling, buzzing, pinching, burning, and/or sharp jabbing stabbing pain in the feet. Nerve pain from diabetic peripheral neuropathy can be severe, constant, and difficult to treat. Current therapies include an array of over-the-counter and prescription medications or alternative treatment options such as injections or patches of local anesthetics; surgical destruction of nerves; implantation of a device to relieve pain; transcutaneous electrotherapy (TENS); hand or foot braces and orthopedic shoes.

Low Level Laser Therapy (LLLT) communicates information to the receptors on the membrane of the cell and mitochondrion (the enzymatic engine of the cell). This energetic information reaches the cell's DNA, which directly controls cell function. When the cells receive better information, they work better, as do the tissues they comprise, like bones, cartilage, tendons, ligaments, etc. In this way, LLLT promotes the healing and regeneration of damaged tissues, having both local effects on tissue function and also systemic effects carried throughout the body by the blood and acupuncture meridians.

The key basic physiological effects of low level laser light include increased cell membrane polarization and permeability; Adenosine-5-triphosphate (ATP) production and respiratory chain activity; enzyme activity; collagen and epithelial production; capillary formation; macrophage (immune) activity; analgesic effects due to elevated endorphin production, electrolytic nerve blockage, and improved blood and lymph flow; anti-inflammatory effect due to improved circulation and accelerated tissue regeneration; and increased production of antioxidants. Of additional benefit is that light energy from low level lasers will only be absorbed by cells and tissues that are not functioning normally and has no effect on healthy cells.

Therefore, low level laser therapy has the potential benefit of providing an effective means of reducing low back pain that is simple, quick, non-invasive and side-effect free.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older. Significant spontaneous pain of 50 or greater on the 0-100 VAS for the feet overall.
* Existing clinical diagnosis of diabetes induced Peripheral Neuropathy.
* Significant spontaneous foot pain that occurs comparably bilaterally.
* Foot pain is chronic, ongoing for at least 3 months, bilaterally.
* Subject has been on a stable anti-diabetic medication regimen or on no anti-diabetic medication regimen for the prior 30 days.
* Subject has not used or is willing to abstain from using analgesics within 7 days prior to study start.
* Subject has been on a stable dosage of antidepressants for at least 90 days prior to study start and is willing and able to maintain that stable dosage throughout study participation OR subject has not used or is willing to abstain from using antidepressants for 30 days prior to study start.
* Subject has been on a stable dosage of any of Neurontin, Lyrica, Tramadol and Opioid medicines such as Ultram and Ultracet for at least 90 days prior to study start and is willing and able to maintain that stable dosage throughout study participation OR subject has not used or is willing to abstain from using any of the these medications for 30 days prior to study start.
* Subject has not received or is willing to abstain from receiving any injections of local anesthetics such as lidocaine within 30 days prior to study start.
* Subject is able and willing to take over-the-counter Regular Strength Tylenol tablets to manage pain, as needed, throughout the study.
* Subject is willing and able to refrain from consuming any over-the-counter and/or prescription medications including muscle relaxants and/or herbal supplements and/or recreational and medical drugs including cannabis intended for the relief of pain and/or inflammation throughout study participation, except for the study-specific pain relief medication of over-the-counter Tylenol.
* Subject is willing and able to refrain from engaging in any non-study procedure therapies for the management of foot pain throughout the study, including conventional therapies such as physical therapy, occupational therapy and hot or cold packs, as well as alternative therapies such as chiropractic care and acupuncture.
* Can communicate fluently in English and can read and write English sufficiently to comply with the study procedures and complete the information in the Subject Diary.

Exclusion Criteria:

* Subject's foot pain is undiagnosed, or has been diagnosed as being other than, or in addition to, diabetes induced Peripheral Neuropathy.
* Subject's foot pain is unilateral or notably different between the two feet.
* Serious organ disease or other serious primary disease merger.
* Diabetes ketosis, ketoacidosis or severe infection within the past two weeks.
* Current, active chronic pain disease: chronic fatigue syndrome, fibromyalgia, endometriosis, inflammatory bowel disease, interstitial cystitis, peripheral vascular disease.
* Cancer or treatment for cancer in the past 6 months.
* Surgical intervention to treat diabetic peripheral neuropathy foot pain, including implantation of a pain relief device.
* Active infection, wound, or other external trauma to the areas to be treated with the laser.
* Medical, physical, or other contraindications for, or sensitivity to, light therapy.
* Pregnant, breast feeding, or planning pregnancy prior to the end of study participation.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.
* Any condition or other variable that in the opinion of the investigator may confound or interfere with the evaluation of the effectiveness of the investigational treatment or otherwise render the subject unable to comply with the requirements of the study protocol.
* Involvement in litigation and/or receiving disability benefits related in any way to the parameters of the study.
* Participation in a clinical study or other type of research in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Franco, DPM, Principal Investigator
Locations (4):
- United States (4):
  - Arizona Institute of Footcare Physicians, Mesa, Arizona
  - Jeffrey Kleis, DPM, Costa Mesa, California
  - Hialeah Hospital Medical Plaza, Hialeah, Florida
  - Jordan Steinberg, DPM, Florham Park, New Jersey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia FX-635 | Placebo Laser
Started | 11 | 7
Completed | 11 | 6
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia FX-635 | Placebo Laser | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (3) | 67.3 (8.80) | 65.6 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Participants With a 30% or Greater Change in Visual Analog Scale (VAS) Pain Scores
Description: The Visual Analog Scale (VAS) assesses level or degree of pain. It is a horizontal line anchored on the left by the label '0: no pain at all' and on the right by the label '100: worst pain imaginable'. The subject marks a location on the 0-100 line that appears to represent any level of pain he or she is experiencing at that time. This marking is measured with a 0 to 100 mm ruler and the number recorded. For the primary study outcome, the percent change in the VAS pain score recorded at baseline and endpoint is calculated for each subject. Individual subject success is a 30% or greater change in VAS pain scores. A negative (-) percent change indicates a decrease in pain level and is positive for individual subject success. A positive (+) percent change indicates an increase in pain level and is negative for individual subject success. Overall study success is defined as a 35% or greater difference between the proportion of individual successes in each treatment group.
Time Frame: Baseline and 6 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia FX-635 | Placebo Laser
Number analyzed (Participants) | 11 | 6
participants | 4 | 1

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Erchonia FX-635 | Placebo Laser
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6
Other Adverse Events (participants affected / at risk) | 0/11 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT04006392/Prot_SAP_000.pdf